CLINICAL TRIAL: NCT00420173
Title: Interdisciplinary Study Group of Lupus Erythematosus
Brief Title: Interdisciplinary Study Group of Lupus Erythematosus (ISGLE)
Status: Completed | Type: Observational
Sponsor: European Society of Cutaneous Lupus Erythematosus e.V. (Other)
Responsible Party: Principal Investigator, Prof. Dr. Annegret Kuhn, Professor, Kuhn, Annegret
Other Study IDs: 2742-1
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Cutaneous Lupus Erythematosus
Keywords: cutaneous lupus erythematosus; standardized evaluation; core set questionnaire; epidemiological data; laboratory features
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with CLE
  Interventions: Procedure: Laboratory analysis

INTERVENTIONS:
Procedure: Laboratory analysis — blood withdrawal

SUMMARY:
Cutaneous lupus erythematosus (CLE) is a disease with a wide spectrum of clinical manifestations and a variable prognosis. The aim of this study is to create a standardized evaluation of the different subtypes of this disease in order to receive an overview of the spectrum of clinical and laboratory features as well as the therapeutic strategies for patients with CLE.

DETAILED DESCRIPTION:
Methods: A core set questionnaire has been developed in the course of the "European Society of Cutaneous Lupus Erythematosus (EUSCLE)", and a total of 40 patients (32 females, 8 males) in two centres, Germany and Sweden, were included in this study. Results: CLE was diagnosed in 39 individuals (5 with acute CLE, 10 with subacute CLE, 13 with chronic CLE, and 18 with intermittent CLE) and one individual presented with a systemic manifestation of the disease. Furthermore, disease onset and duration as well as activity and damage of skin lesions using a modified CLASI were examined. Interestingly, 75% of the patients with CLE showed a positive history of photosensitivity, but only 62.5% exhibited characteristic lesions after standardized phototesting. Laboratory analysis revealed positive antinuclear antibodies in 50% of the patients, positive anti-Ro/SSA in 12 and positive anti-La/SSB antibodies in 8 cases. The predominantly used treatments included sunscreens (38 patients), topical steroids (31 patients), topical calcineurin inhibitors (12 patients), chloroquine (19 patients), hydroxychloroquine (11 patients), and systemic steroids (12 patients). Conclusions: The new core set questionnaire enables the clinician to characterize the different skin manifestations involved in CLE and to evaluate disease activity and reasonable treatment modalities. Furthermore, epidemiological data and laboratory features can be assessed for the various subtypes. In the future, this standardized evaluation might lead to the development of diagnostic guidelines and evidence based therapeutic strategies thus improving quality of care for patients with CLE.

ELIGIBILITY:
Inclusion Criteria:

* cutaneous lupus erythematosus confirmed by histological analysis
* photoprovocation-test performed in advance
* written informed consent available prior to any procedures

Exclusion Criteria:

* patients with conditions that are contrary to the above mentioned criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cutaneous lupus erythematosus
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2004-09; Primary Completion 2005-07 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Kuhn, MD, Principal Investigator — Universität Münster
Locations (1):
- University of Muenster, Department of Dermatology, Münster, North Rhine-Westphalia, Germany